CLINICAL TRIAL: NCT05647057
Title: Optimization of Prime Fluid Strategy to Preserve Microcirculatory Perfusion During Cardiac Surgery With Cardiopulmonary Bypass
Brief Title: CPB Prime Fluid Strategies to Preserve Mcirocirculatory Perfusion
Acronym: PRIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Alexander B.A. Vonk, Cardiothoracic surgeon, Principle Investigator, doctor., Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL82500.029.22, part I
Record Dates: First submitted 2022-11-09; First posted 2022-12-12 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Endothelial Dysfunction; Hemolysis; Fluid Overload
Keywords: Microcirculation; Cardiopulmonary bypass; Colloid oncotic pressure; Hemodilution; Hemolysis
MeSH Terms: conditions — Hemolysis; Edema

STUDY DESIGN:
Intervention Model Description: In two consecutive randomized controlled trials, the investigators study the effect of prime fluid strategies on perfused vessel density (part I) and the effect of additional albumin during cardiopulmonary bypass compared with ringers on perfused vessel density (part II).
  In this study part (I), the effect of prime fluid strategies on perfused vessel density.
  A single centre, double-blind randomized trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: gelofusine + ringers (Active Comparator): Prime fluid strategy containing gelofusine and ringers
  Interventions: Combination Product: A: gelofusine + ringers
- B: albumin + ringers (Active Comparator): Prime fluid strategy containing albumin and ringers
  Interventions: Combination Product: B: albumine + ringers
- C: ringers + retrograde autologous priming (Active Comparator): Prime fluid strategy containing ringers combined with retrograde autologous priming
  Interventions: Combination Product: C: ringers + retrograde autologous priming

INTERVENTIONS:
Combination Product: A: gelofusine + ringers — 750 milliliter (mL) modified fluid gelatin (Braun Melsungen, Germany), 650 mL Ringer's solution (Baxter, Utrecht, Netherlands) and 100 mL mannitol (15%, Baxter, Utrecht, Netherlands)
  Arms: A: gelofusine + ringers
Combination Product: B: albumine + ringers — 200 mL human albumin (20%, Sanquin, Amsterdam, Netherlands), 1200 mL Ringer's solution (Baxter, Utrecht, Netherlands) and 100 mL mannitol (15%, Baxter, Utrecht, Netherlands)
  Arms: B: albumin + ringers
Combination Product: C: ringers + retrograde autologous priming — 1400 mL Ringer's solution (Baxter, Utrecht, Netherlands) and 100 mL mannitol (15%, Baxter, Utrecht, Netherlands) with retrograde autologous priming.
  Retrograde autologous priming (RAP) is applied using clinical parameters such as Central Venous Pressure, Mean Arterial Pressure (MAP), and intra cardiac filling pressure based on Trans Esophageal Echo as guidance to the amount of fluid displaced. RAP is applied to a maximum volume of 475 mL provided that systolic blood pressure will remain >90 millimeter of mercury (mmHg). Phenylephrine can be administered up to 200 mcg to keep the system hemodynamics stable during RAP. In case of a body surface area <1.7m2, a maximum volume of 375 mL is desired. Once the desired amount of prime is displaced, the transfusion bag is clamped and CPB is started. If additional fluids are needed during CPB to maintain optimal perfusion, the displaced prime is used prior to the vasoplegia protocol.
  Arms: C: ringers + retrograde autologous priming

SUMMARY:
Acute microcirculatory perfusion disturbances is common in critical illness and associated with higher morbidity and mortality. Recent findings by the investigators' group showed that microcirculatory perfusion is disturbed during cardiac surgery with cardiopulmonary bypass (CPB) and remain disturbed up to 72 (seventy two) hours after surgery. A cardiopulmonary bypass is a machine which takes over heart and lung function, during the procedure. The disturbed microcirculation is associated with organ dysfunction induced by cardiac surgery using CPB, which is frequently seen (up to 42%, forty two percent) and results in a six-fold increase in mortality rate. The underlying cause of disturbed microcirculation is a higher endothelial permeability and vascular leakage and are a consequence of systemic inflammation, hemodilution (dilution of blood), hypothermia and hemolysis (breakdown of red blood cells). To gain the knowledge regarding disturbed microcirculation the investigators previously showed that hemodilution attributes to this disturbed perfusion. Hemodilution lowers colloid oncotic pressure (COP). Also, COP is affected by free hemoglobin, which increases with hemolysis and attributes to a disturbed microcirculation following CPB. This is interesting, as to the best of our knowledge, the effect of minimizing hemodilution and hemolysis during cardiac surgery on the microcirculatory perfusion has never been investigated, but could be the key factor in reducing organ dysfunction.

DETAILED DESCRIPTION:
In this project the investigators focus on reducing microcirculatory perfusion disturbances by exploring therapeutic approaches with different prime fluid strategies, by acting on COP (part I) and free hemoglobin scavenging with human albumin (part II).

In part I, patients undergoing elective coronary artery bypass graft (CABG) surgery with cardiopulmonary bypass will be randomized in three groups receiving different prime fluid strategies. The study endpoint is the reduction in functional capillary density during the perioperative period. Sublingual microcirculatory measurements and blood sampling will take place after induction of anesthesia, during and after surgery to determine microcirculatory perfusion and parameters for hemodilution, hemolysis, COP, markers for endothelial damage and glycocalyx shedding. Measurements start on the day of surgery and end one day after surgery.

In part II, participants will be randomized in two groups receiving the first dose directly after aortic cross clamping and blood cardioplegia administration, and the second dose after the third blood cardioplegia administration (± 30 min after the first dose).The most optimal prime fluid in order to preserve microcirculatory perfusion from study one, will be used as prime fluid in the second study. Microcirculatory perfusion parameters will be measured at time points comparable with study one. Blood samples are taken to determine markers for hemodilution, hemolysis, COP and endothelial damage and glycocalyx shedding. For part II see trial registration: PRIME, part II.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects
* Informed consent
* Elective coronary artery bypass surgery with cardiopulmonary bypass

Exclusion Criteria:

* Emergency operations
* Re-operation
* Elective thoracic aortic surgery
* Elective valve surgery
* The use of crystalloid cardioplegia
* Combined procedure CABG and valve surgery
* Known allergy for human albumin or gelofusine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
Perfused vessel density (PVD, mm mm-²) | T1: within 5-10 minutes after induction of anesthesia
  reflecting microcirculatory diffusion capacity
Perfused vessel density (PVD, mm mm-²) | T2 within 5-10 minutes after aortic cross clamping
  reflecting microcirculatory diffusion capacity
Perfused vessel density (PVD, mm mm-²) | T3 within 5-10 minutes after weaning from cardiopulmonary bypass
  reflecting microcirculatory diffusion capacity
Perfused vessel density (PVD, mm mm-²) | T4 within 15-30 min after arrival on the intensive care unit
  reflecting microcirculatory diffusion capacity
Perfused vessel density (PVD, mm mm-²) | T5 twenty four (24) hours after arrival on the intensive care unit
  reflecting microcirculatory diffusion capacity

SECONDARY OUTCOMES:
Colloid oncotic pressure (COP, mmHg) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  colloid oncotic pressure in plasma
albumin (g L-¹) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  concentration of albumin in plasma
hemolysis index (H-index) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  the grade of hemolysis in plasma
haptoglobin (g L-¹) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  concentration of haptoglobin in plasma
syndecan-1 (ng/ml) | T1, 5-10 min after induction of anesthesia; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Concentration of syndecan-1 in plasma
heparan sulphate (ng/ml) | T1, 5-10 min after induction of anesthesia; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  concentration of heparan sulphate in plasma
hemoglobin (Hb, mmol L-¹) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  concentration of hemoglobin in serum
hematocrit (Ht, L L-¹) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  hematocrit in serum
perioperative use of packed red blood cells (PRBCs, mL) | Intraoperative during cardiac surgery, postoperative period up to 24 hours postoperative
  amount of packed red blood cells
fluid balance (mL) | Intraoperative during cardiac surgery, postoperative period up to 24 hours postoperative
  fluid balance
fluid requirements (mL) | Intraoperative during cardiac surgery, postoperative period up to 24 hours postoperative
  Amount of fluids required
Total vessel density (TVD, mm mm-²) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  density of capillaries reflecting the functional state of the microcirculatory diffusion capacity
Proportion of perfused vessels (PPV, %) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  reflecting the aspect of heterogeneity of microcirculatory perfusion
Heterogeneity index | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  reflecting the aspect of heterogeneity of microcirculatory perfusion
Thrombomodulin (ng mL-¹) | T1, 5-10 min after induction of anesthesia; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Thrombomodulin concentration in plasma
Angiopoietin-2 (ng mL-¹) | T1, 5-10 min after induction of anesthesia; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Angiopoietin-2 concentration in plasma
Interleukin-6 (ng mL-¹) | T1, 5-10 min after induction of anesthesia; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Interleukin-6 concentration in plasma
Tumor necrosis factor (TNF-alpha, ng mL-¹) | T1, 5-10 min after induction of anesthesia; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  TNF-alpha concentration in plasma
Neutrophil gelatinase associated lipocalin (NGAL, ng mL-¹) | T1, 5-10 min after induction of anesthesia; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  NGAL concentration in plasma
Magnesium (mmol L-¹) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Magnesium concentration in plasma
Phosphate (mmol L-¹) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Phosphate concentration in plasma
Oxygen delivery (mL min-¹) | During cardiopulmonary bypass
  Oxygen delivery
Microvascular Flow Index | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Microvascular Flow Index, semi-quantitative assessment of the average red blood cell velocity per quadrant
De Backer-score | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  De Backer-score, proxy of total vessel density

OTHER OUTCOMES:
Age | Preoperative
  Age in years
Gender | Preoperative
  Gender (male/female)
Body Surface Area (BSA) | Preoperative
  BSA in m2
Smoking | Preoperative
  Medical history of smoking (yes/no)
Diabetes on medication | Preoperative
  Medical history of diabetes on medication (yes/no)
Comorbidities | Preoperative
  Other comorbidities in medical history (yes/no)
EuroSCORE II | Preoperative
  The European System for Cardiac Operative Risk Evaluation (EuroSCORE) II predicts risk of in-hospital mortality after cardiac surgery.
CPB time (min) | intraoperative
  Cardiopulmonary bypass time in minutes
Aortic cross clamping time (AoX time, min) | intraoperative
  Aortic cross clamping time in minutes
heparin (IU) | intraoperative
  Dosing of heparin in international units
protamin (mg) | intraoperative
  dosing of protamin
Activated Clotting Time (ACT, min) | intraoperative
  ACT in minutes
Temperature (celsius) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Temperature in celsius
Oxygen saturation (Sat, %) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Oxygen saturation in %
Urine production (ml) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Urine production
Blood pressure (mmHg) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Blood pressure (mmHg)
Noradrenaline infusion | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Noradrenaline infusion (mcg/kg/min)
Phenylephrine | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Phenylephrine (mcg)
Vasopressin (IU/min) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Vasopressin (IU/min)
Methylene Blue (mg) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Methylene blue (mg)
Lactate (mmol/L) | T1, 5-10 min after induction of anesthesia; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Serum lactate
Creatinin levels (umol/L) | T1, 5-10 min after induction of anesthesia; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  serum creatinin level
estimated glomerular filtration rate (eGFR, ml/min/1,73 m2) | T1, 5-10 min after induction of anesthesia; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  estimated glomerular filtration rate
Blood product use | Intraoperative and up to 24 hours postoperative
  Blood product use (ml)
Blood loss (ml) | T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit
  Blood loss
Duration of mechanical ventilation (hours) | Postoperative until 30 days postoperative
  Duration of mechanical ventilation (hours)
ICU stay (hours) | Postoperative until 30 days postoperative
  ICU stay (hours)
Hospital stay (days) | Postoperative until 30 days postoperative
  Days until hospital discharge (days)
Acute Kidney injury (AKI) | Postoperative until 30 days postoperative
  Acute kidney injury (yes/no)
Respiratory failure | Postoperative until 30 days postoperative
  Respiratory failure (yes/no)
Pneumonia | Postoperative until 30 days postoperative
  Pneumonia (yes/no)
non-preexisting atrial fibrillation | Postoperative until 30 days postoperative
  non-preexisting atrial fibrillation (yes/no)
re-do surgery | Postoperative until 30 days postoperative
  re-do surgery (yes/no)
Extra corporeal membrane oxygenation (ECMO) | Postoperative until 30 days postoperative
  Extra corporeal membrane oxygenation (yes/no)
Mortality | Postoperative until 30 days postoperative
  In-hospital mortality (yes/no)
Sodium (mmol/L) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Serum sodium
Potassium (mmol/L) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Serum potassium
Calcium (mmol/L) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Serum calcium
Chloride (mmol/L) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Serum chloride
Bicarbonate (mmol/L) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Serum bicarbonate
CO2 (kPa) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Carbon dioxide pressure in plasma
O2 (kPa) | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Oxygen pressure in plasma
pH | T1, 5-10 min after induction of anesthesia; T2, 5-10 min after aortic cross clamping; T3, 5-10 min after weaning from cardiopulmonary bypass; T4, 15-30 min after arrival on the intensive care unit; T5, 24 hours after arrival on the intensive care unit.
  Measurement of hydrogen ions in plasma

CONTACTS AND LOCATIONS:
Overall Officials: A.B.A. Vonk, MD, PhD, Principal Investigator — Cardiothoracic surgeon
Locations (1):
- Amsterdam UMC, AMC location, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: SAP, Analytic Code
Time Frame: Upon request

REFERENCES:
- [Derived] Beukers AM, Bulte CSE, Bosch RJ, Eberl S, van den Brom CE, Loer SA, Vonk ABA. Optimization of cardiopulmonary bypass prime fluid to preserve microcirculatory perfusion during on-pump coronary artery bypass graft surgery: PRIME study protocol for a double-blind randomized trial. Trials. 2024 Mar 26;25(1):219. doi: 10.1186/s13063-024-08053-5. PMID 38532434

DOCUMENTS (1):
  • Study Protocol: Explanation of Randomization process (2025-03-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT05647057/Prot_000.pdf